CLINICAL TRIAL: NCT01795937
Title: Investigation of Interactions Between Faldaprevir, Itraconazole, Atorvastatin and Rosuvastatin in Healthy Male and Female Subjects (Open-label, Fixed-sequence)
Brief Title: Investigation of Interactions Between Faldaprevir, Itraconazole, Atorvastatin and Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1220.61; 2012-005518-20 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-02-20; First posted 2013-02-21 (Estimated); Results first posted 2015-08-03 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole; Atorvastatin; faldaprevir; Rosuvastatin Calcium

ARMS (2):
- Part 1: Faldaprevir + Itraconazole (Experimental): Interaction of Faldaprevir and Itraconazole
  Interventions: Drug: Itraconazole; Drug: Faldaprevir
- Part 2:Faldaprevir+Rosuvastatin+Atorvast (Experimental): Interaction of Faldaprevir, Rosuvastatin and Atorvastatin
  Interventions: Drug: Atorvastatin; Drug: Faldaprevir; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Itraconazole — twice daily
  Arms: Part 1: Faldaprevir + Itraconazole
Drug: Atorvastatin — single dose
  Arms: Part 2:Faldaprevir+Rosuvastatin+Atorvast
Drug: Faldaprevir — once daily
  Arms: Part 2:Faldaprevir+Rosuvastatin+Atorvast
Drug: Rosuvastatin — single dose
  Arms: Part 2:Faldaprevir+Rosuvastatin+Atorvast
Drug: Faldaprevir — once daily
  Arms: Part 1: Faldaprevir + Itraconazole

SUMMARY:
To investigate the effect of steady-state itraconazole on the pharmacokinetics of steady-state of faldaprevir and the effect of steady-state of faldaprevir on the single-dose pharmacokinetics of atorvastatin as well as the effect of steady-state of faldaprevir on the single-dose pharmacokinetics of rosuvastatin

ELIGIBILITY:
Inclusion criteria:

1. Healthy male and female subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2013-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1220.61.1 Boehringer Ingelheim Investigational Site, Ingelheim, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Sequence A_B (Itraconazole Part): The itraconazole part (interaction of steady state faldaprevir with itraconazole) of this trial was done open-label with a fixed-sequence, 2-period design; performed independently from the statins part.
  Treatment A: Faldaprevir (120 mg) was given twice daily on Day -5 and once daily from Day -4 to Day 1 (6 days in total).
  Treatment B: Faldaprevir (120 mg) was given once daily from Day -3 to Day 1 (4 days). In addition, itraconazole (200 mg) was given twice daily on Day -3 and once daily from Day -2 to Day 1 (4 days in total).
  Treatment A directly preceded treatment B, without an intermittent washout period.
  Oral administration with 240 mL water.
- Treatment Sequence C_D (Statins Part): The statins part (interaction of multiple dose faldaprevir with either atorvastatin or rosuvastatin) was done open-label with a fixed-sequence, 2-period design; performed independently from the itraconazole part.
  Treatment C: Atorvastatin (10 mg) was given as a single dose on Day 1.
  Treatment D: Faldaprevir (240 mg) was given twice daily on Day -5 and once daily from Day -4 to Day 2 (7 days in total). In addition, atorvastatin (10 mg) was given as a single dose on Day 1.
  Treatment C preceded treatment D.
  Oral administration with 240 mL water.
- Treatment Sequence E_F (Statins Part): The statins part (interaction of multiple dose faldaprevir with either atorvastatin or rosuvastatin) was done open-label with a fixed-sequence, 2-period design; performed independently from the itraconazole part.
  Treatment E: Rosuvastatin (10 mg) was given as a single dose on Day 1.
  Treatment F: Faldaprevir (240 mg) was given twice daily on Day -5 and once daily from Day -4 to Day 2 (7 days in total). In addition, rosuvastatin (10 mg) was given as a single dose on Day 1.
  Treatment E preceded treatment F.
  Oral administration with 240 mL water.
Period: Overall Study
Arm/Group | Treatment Sequence A_B (Itraconazole Part) | Treatment Sequence C_D (Statins Part) | Treatment Sequence E_F (Statins Part)
Started | 18 | 16 | 17
Completed | 17 | 15 | 17
Not Completed | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The itraconazole part of this trial was done open-label with a fixed-sequence, 2-period design (treatment seq. A_B).
  The statins part was done open-label with a fixed-sequence, 2-period design. Subjects in the statins part were assigned to 1 of the 2 possible treatment sequences: treatment seq. C_D or E_F.
  Both parts were performed independently.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence A_B (Itraconazole Part) | Treatment Sequence C_D (Statins Part) | Treatment Sequence E_F (Statins Part) | Total
Number analyzed (Participants) | 18 | 16 | 17 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (6.8) | 40.0 (8.3) | 38.1 (7.4) | 39.3 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 10 | 22
  Male | 10 | 12 | 7 | 29

OUTCOME MEASURES:

1. Primary Outcome: AUCτ,ss (Itraconazole Part)
Description: Area under the concentration-time curve of the analyte in plasma at steady state over the dosing interval τ (AUCτ,ss) of faldaprevir. Outcome measure for the itraconazole part (treatment sequence A_B) of this trial. The measured values show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: -1:30, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 11:00, 12:00 h (hours) after administration of faldaprevir on Day 1 of both periods
Population: pharmacokinetic (PK) set of the itraconazole part of this trial. The PK set included all treated subjects of the itraconazole part that provided at least 1 observation for at least 1 primary endpoint without important protocal violations with respect to the statistical evaluation of the PK endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Faldaprevir: Faldaprevir 120 mg once daily from Day -4 to Day 1 with a 120 mg twice daily loading dose on Day -5 (6 days in total).
  Treatment A.
- Faldaprevir+Itraconazole: Faldaprevir 120 mg once daily from Day -3 to Day 1 + itraconazole 200 mg twice daily on Day -3 and once daily from Day -2 to Day 1 (4 days in total).
  Treatment B.
Arm/Group | Faldaprevir | Faldaprevir+Itraconazole
Number analyzed (Participants) | 17 | 17
ng*h/mL | 29900 (62.8) | 59500 (53.8)
Statistical Analysis 1: Comparison: Faldaprevir vs Faldaprevir+Itraconazole; Relative bioavailability comparison faldaprevir+itraconazole : faldaprevir; Test type: Non-Inferiority or Equivalence — Investigation of relative bioavailability (no formal testing); ANOVA; ANOVA with fixed effect for treatment and random effect for subject; Geometric Mean Ratio = 198.55, 90% CI 2-sided [182.43 to 216.09], Standard Deviation 14.2 — The standard deviation is actually the geometric coefficient of variation

2. Primary Outcome: Cmax,ss (Itraconazole Part)
Description: Maximum measured concentration of the analyte in plasma at steady state over the dosing interval (Cmax,ss) of faldaprevir. Outcome measure for the itraconazole part (Treatment sequence A_B) of this trial.
  The measured values show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: -1:30, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 11:00, 12:00 h after administration of faldaprevir on Day 1 of both periods.
Population: PK set of the itraconazole part of this trial.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Faldaprevir | Faldaprevir+Itraconazole
Number analyzed (Participants) | 17 | 17
ng/mL | 2780 (61.0) | 5030 (49.1)
Statistical Analysis 1: Comparison: Faldaprevir vs Faldaprevir+Itraconazole; Relative bioavailability comparison faldaprevir+itraconazole : faldaprevir; Test type: Non-Inferiority or Equivalence — Investigation of relative bioavailability (no formal testing); ANOVA; ANOVA with fixed effect for treatment and random effect for subject; Geometric Mean Ratio = 180.63, 90% CI 2-sided [165.68 to 196.93], Standard Deviation 14.5 — The standard deviation is actually the geometric coefficient of variation

3. Primary Outcome: AUC0-∞ of Atorvastatin (Statins Part)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) of atorvastatin after single dose administration. Outcome measure for the statins part of this trial, treatment sequence C_D.
  The measured values show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: -1:30, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 11:00, 12:00, 24:00, 36:00, 48:00, 60:00 h after administration of atorvastatin on Day 1 of both periods.
Population: PK set of the statins part and assigned to atorvastatin (treatment sequence C_D).
  Pharmacokinetic set (PK set): all treated subjects of the statins part that provided at least 1 observation for at least 1 primary endpoint without important protocol violations with respect to the statistical evaluation of the pharmacokinetic endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Atorvastatin: Atorvastatin (10 mg) was given as a single dose on Day 1.
  Treatment C.
- Atorvastatin+Faldaprevir: Faldaprevir (240 mg) was given twice daily on Day -5 and once daily from Day -4 to Day 2 (7 days in total). In addition, atorvastatin (10 mg) was given as a single dose on Day 1.
  Treatment D.
Arm/Group | Atorvastatin | Atorvastatin+Faldaprevir
Number analyzed (Participants) | 16 | 15
ng*h/mL | 13.7 (51.5) | 129.0 (43.7)
Statistical Analysis 1: Comparison: Atorvastatin vs Atorvastatin+Faldaprevir; Relative bioavailability comparison atorvastatin+faldaprevir : atorvastatin; Test type: Non-Inferiority or Equivalence — Investigation of relative bioavailability (no formal testing); ANOVA; ANOVA with fixed effect for treatment and random effect for subject; Geometric Mean Ratio = 946.45, 90% CI 2-sided [797.61 to 1123.07], Standard Deviation 27.3 — The standard deviation is actually the geometric coefficient of variation

4. Primary Outcome: Cmax of Atorvastatin (Statins Part)
Description: Maximum measured concentration of the analyte in plasma of atorvastatin (Cmax). Outcome measure for the statins part of this trial, treatment sequence C_D.
  The measured values show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: as for outcome 3
Population: PK set of the statins part and assigned to atorvastatin (treatment sequence C_D).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Atorvastatin | Atorvastatin+Faldaprevir
Number analyzed (Participants) | 16 | 15
ng/mL | 0.94 (35.2) | 31.10 (52.5)
Statistical Analysis 1: Comparison: Atorvastatin vs Atorvastatin+Faldaprevir; Relative bioavailability comparison atorvastatin+faldaprevir : atorvastatin; Test type: Non-Inferiority or Equivalence — Investigation of relative bioavailability (no formal testing); ANOVA; ANOVA with fixed effect for treatment and random effect for subject; Geometric Mean Ratio = 3372.72, 90% CI 2-sided [2961.95 to 3840.47], Standard Deviation 20.5 — The standard deviation is actually the geometric coefficient of variation

5. Secondary Outcome: AUCτ,ss of Faldaprevir (Statins Part)
Description: Area under the concentration-time curve of the analyte in plasma at steady state over the dosing interval τ (AUCτ,ss) of faldaprevir. Outcome measure for the statins part of this trial, treatment sequences C_D and E_F.
Time Frame: -1:30, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 11:00, 12:00, 24:00, 36:00, 48:00, 60:00 h after administration of rosuvastatin/atorvastatin on Day 1 of the second periods of each treatment sequence.
Population: PK set of the statins part.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Rosuvastatin+Faldaprevir: Faldaprevir (240 mg) was given twice daily on Day -5 and once daily from Day -4 to Day 2 (7 days in total). In addition, rosuvastatin (10 mg) was given as a single dose on Day 1.
  Treatment F.
Arm/Group | Atorvastatin+Faldaprevir | Rosuvastatin+Faldaprevir
Number analyzed (Participants) | 15 | 17
ng*h/mL | 145000 (34.3) | 136000 (43.9)

6. Secondary Outcome: Cmax,ss of Faldaprevir (Statins Part)
Description: Maximum measured concentration of the analyte in plasma at steady state over the dosing interval (Cmax,ss) of faldaprevir. Outcome measure for the statins part of this trial, treatment sequences C_D and E_F.
Time Frame: as for outcome 5
Population: PK set of the statins part.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Atorvastatin+Faldaprevir | Rosuvastatin+Faldaprevir
Number analyzed (Participants) | 15 | 17
ng/mL | 12900 (27.8) | 12200 (36.8)

7. Secondary Outcome: AUC0-tz of Atorvastatin
Description: Area under the plasma concentration-time curve of the analyte over the time interval from 0 to the time tz of the last measurable concentration (AUC0-tz) of atorvastatin. Outcome measure for the statins part of this trial, treatment sequence C_D.
  The measured values show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: as for outcome 3
Population: PK set of the statins part and assigned to atorvastatin (treatment sequence C_D).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Atorvastatin | Atorvastatin+Faldaprevir
Number analyzed (Participants) | 16 | 15
ng*h/mL | 9.5 (40.2) | 129.6 (44.9)
Statistical Analysis 1: Comparison: Atorvastatin vs Atorvastatin+Faldaprevir; Relative bioavailability comparison atorvastatin+faldaprevir : atorvastatin; Test type: Non-Inferiority or Equivalence — Investigation of relative bioavailability (no formal testing); ANOVA; ANOVA with fixed effect for treatment and random effect for subject; Geometric Mean Ratio = 1358.91, 90% CI 2-sided [1224.32 to 1508.29], Standard Deviation 16.4 — The standard deviation is actually the geometric coefficient of variation

8. Primary Outcome: AUC0-∞ of Rosuvastatin (Statins Part)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) of rosuvastatin after single dose administration of rosuvastatin. Outcome measure for the statins part of this trial, treatment sequence E_F.
  The measured values show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: -1:30, 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 11:00, 12:00, 24:00, 36:00, 48:00, 60:00 h after administration of rosuvastatin on Day 1 of both periods
Population: PK set of the statins part and assigned to rosuvastatin (treatment sequence E_F).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Rosuvastatin: Rosuvastatin (10 mg) was given as a single dose on Day 1.
  Treatment E.
Arm/Group | Rosuvastatin | Rosuvastatin+Faldaprevir
Number analyzed (Participants) | 17 | 17
ng*h/mL | 24.9 (49.3) | 365.0 (28.6)
Statistical Analysis 1: Comparison: Rosuvastatin vs Rosuvastatin+Faldaprevir; Relative bioavailability comparison rosuvastatin+faldaprevir : rosuvastatin; Test type: Non-Inferiority or Equivalence — Investigation of relative bioavailability (no formal testing); ANOVA; ANOVA with fixed effect for treatment and random effect for subject; Geometric Mean Ratio = 1466.35, 90% CI 2-sided [1277.62 to 1682.95], Standard Deviation 23.3 — The standard deviation is actually the geometric coefficient of variation

9. Primary Outcome: Cmax of Rosuvastatin
Description: Maximum measured concentration of the analyte in plasma of rosuvastatin (Cmax). Outcome measure for the statins part of this trial, treatment sequence E_F.
  The measured values show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: as for outcome 8
Population: PK set of the statins part and assigned to rosuvastatin (treatment sequence E_F).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Rosuvastatin | Rosuvastatin+Faldaprevir
Number analyzed (Participants) | 17 | 17
ng/mL | 2.73 (53.0) | 89.6 (33.2)
Statistical Analysis 1: Comparison: Rosuvastatin vs Rosuvastatin+Faldaprevir; Relative bioavailability comparison rosuvastatin+faldaprevir : rosuvastatin; Test type: Non-Inferiority or Equivalence — Investigation of relative bioavailability (no formal testing); ANOVA; ANOVA with fixed effect for treatment and random effect for subject; Geometric Mean Ratio = 3288.70, 90% CI 2-sided [2782.04 to 3887.63], Standard Deviation 28.5 — The standard deviation is actually the geometric coefficient of variation

10. Secondary Outcome: AUC0-tz of Rosuvastatin
Description: Area under the plasma concentration-time curve of the analyte over the time interval from 0 to the time tz of the last measurable concentration (AUC0-tz) of rosuvastatin. Outcome measure for the statins part of this trial, treatment sequence E_F.
  The measured values show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: as for outcome 8
Population: PK set of the statins part and assigned to rosuvastatin (treatment sequence E_F).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Rosuvastatin | Rosuvastatin+Faldaprevir
Number analyzed (Participants) | 17 | 17
ng*h/mL | 21.5 (48.0) | 361.0 (28.8)
Statistical Analysis 1: Comparison: Rosuvastatin vs Rosuvastatin+Faldaprevir; Relative bioavailability comparison rosuvastatin+faldaprevir : rosuvastatin; Test type: Non-Inferiority or Equivalence — Investigation of relative bioavailability (no formal testing); ANOVA; ANOVA with fixed effect for treatment and random effect for subject; Geometric Mean Ratio = 1678.23, 90% CI 2-sided [1468.52 to 1917.89], Standard Deviation 22.6 — The standard deviation is actually the geometric coefficient of variation

ADVERSE EVENTS:
Time Frame: Adverse events were to be recorded from screening until the end-of-trial examination. Itraconazole part: up to 25 days. Statins part: up to 33 days.
Description: Adverse events were recorded throughout the clinical trial, but were specifically asked for at prespecified time points and additionally whenever the investigator deemed necessary. Subjects were asked to spontaneously report any adverse events as well as the time of onset, end, and intensity.
Groups:
- Faldaprevir (Itraconazole Part): Faldaprevir: 120 mg once daily with a 120 mg twice daily loading dose on Day -5.
  Treatment A.
- Faldaprevir+Itraconazole (Itraconazole Part): Faldaprevir: 120 mg once daily. Itraconazole: 200 mg once daily with a 200 mg twice daily loading dose on Day -3.
  Treatment B.
- Atorvastatin (Statins Part): Atorvastatin: 10 mg was given as a single dose on Day 1.
  Treatment C.
  From the time of the single dose atorvastatin administration in treatment C until the time of the first faldaprevir administration in treatment D or until 1 day after the trial completion date of the respective subject.
- Rosuvastatin (Statins Part): Rosuvastatin: 10 mg was given as a single dose on Day 1.
  Treatment E.
  From the time of the single dose rosuvastatin administration in treatment E until the time of the first faldaprevir administration in treatment F or until 1 day after the trial completion date.
- Faldaprevir (Statins Part): From the time of the first faldaprevir administration in treatment D or F until the combined administration of faldaprevir with atorvastatin or rosuvastatin in treatment D or F, respectively, or until 1 day after the trial completion date.
- Faldaprevir + Atorvastatin (Statins Part): Faldaprevir: 240 mg was given twice daily on Day -5 and once daily from Day -4 to Day 2. Atorvastatin: 10 mg was given as a single dose on Day 1.
  Treatment D.
  From the time of the combined administration of faldaprevir with atorvastatin in treatment D until 1 day after the trial completion date.
- Faldaprevir + Rosuvastatin (Statins Part): Faldaprevir: 240 mg was given twice daily on Day -5 and once daily from Day -4 to Day 2. Rosuvastatin: 10 mg was given as a single dose on Day 1.
  Treatment F.
  From the time of the combined administration of faldaprevir with rosuvastatin in treatment F until 1 day after the trial completion date.
Arm/Group | Faldaprevir (Itraconazole Part) | Faldaprevir+Itraconazole (Itraconazole Part) | Atorvastatin (Statins Part) | Rosuvastatin (Statins Part) | Faldaprevir (Statins Part) | Faldaprevir + Atorvastatin (Statins Part) | Faldaprevir + Rosuvastatin (Statins Part)
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17 | 0/16 | 0/17 | 0/32 | 0/15 | 0/17
Other Adverse Events (participants affected / at risk) | 13/18 | 3/17 | 5/16 | 4/17 | 23/32 | 8/15 | 9/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Faldaprevir (Itraconazole Part) (N=18) | Faldaprevir+Itraconazole (Itraconazole Part) (N=17) | Atorvastatin (Statins Part) (N=16) | Rosuvastatin (Statins Part) (N=17) | Faldaprevir (Statins Part) (N=32) | Faldaprevir + Atorvastatin (Statins Part) (N=15) | Faldaprevir + Rosuvastatin (Statins Part) (N=17)
Nasopharyngitis (Infections and infestations) | 2 | 0 | 1 | 1 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 10 | 0 | 0 | 2 | 3 | 2 | 3
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0 | 2 | 1 | 0
Ocular icterus (Eye disorders) | 1 | 0 | 0 | 0 | 4 | 5 | 3
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 13 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 6 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 6 | 0 | 0 | 1 | 5 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes